CLINICAL TRIAL: NCT05203965
Title: Functional Neuroimaging of Alcoholism Vulnerability: Probing Glutamate and Reward, Using the mGluR5 Inhibitor Mavoglurant
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Godfrey Pearlson, Professor of Psychiatry and of Neuroscience, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HHC-2021-0006; 2P50AA012870-21 (NIH); 2000032425 (Other: Yale IRB)
Record Dates: First submitted 2022-01-05; First posted 2022-01-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Familial Alcoholism Vulnerability
MeSH Terms: interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- FHP; Mavoglurant-Placebo (Experimental): Family History Positive (FHP) for alcoholism will be given a single dose of AFQ056 (200 mg) then placebo in two separate experimental study visits separated by 1 week. Drug and Placebo administered 2 hours prior to the MRI and other measures.
  Interventions: Drug: Mavoglurant (AFQ056); Drug: Placebo
- FHP; Placebo-Mavoglurant (Experimental): Family History Positive (FHP) or alcoholism will be given a single dose of placebo then AFQ056 (200 mg) in two separate experimental study visits separated by 1 week. Drug and Placebo administered 2 hours prior to the MRI and other measures.
  Interventions: Drug: Mavoglurant (AFQ056); Drug: Placebo
- FHN; Mavoglurant-Placebo (Experimental): Family History Negative (FHN) for alcoholism will be given a single dose of AFQ056 (200 mg) then placebo in two separate experimental study visits separated by 1 week. Drug and Placebo administered 2 hours prior to the MRI and other measures.
  Interventions: Drug: Mavoglurant (AFQ056); Drug: Placebo
- FHN; Placebo-Mavoglurant (Experimental): Family History Negative (FHN) for alcoholism will be given a single dose of placebo then AFQ056 (200 mg) in two separate experimental study visits separated by 1 week. Drug and Placebo administered 2 hours prior to the MRI and other measures.
  Interventions: Drug: Mavoglurant (AFQ056); Drug: Placebo

INTERVENTIONS:
Drug: Mavoglurant (AFQ056) — Two 100mg tablets of Mavoglurant will be administered on the morning of one of the two experimental days by a RN or the physician investigator.
Drug: Placebo — Two matching tablets of placebo will be administered on the morning of one of the two experimental days by an RN or the physician investigator.

SUMMARY:
The purpose of this study is to evaluate the role of Mavoglurant in clarifying the neurobiology of alcoholism risk. This is a one-site, randomized, within subjects, counterbalanced double-blind study of a single dose (200mg) of Mavoglurant and placebo.

DETAILED DESCRIPTION:
This project explores the effects of 1 dose of Mavoglurant, an experimental non-competitive antagonist to metabotropic glutamate receptor-5 (mGlur5) developed by Novartis, in a double-blind, randomized, counterbalanced manner on alcoholism risk-relevant tasks. Drug/placebo will be administered on 2 separate visits separated by 1 week. More specifically, this project examines 4 functional MRI tasks related to different aspects of reward and/or impulsivity-related behavior in different contexts, compares the underlying neural circuitry across tasks, and uses a pharmacologic probe of the glutamatergic system to examine N-methyl-D-Aspartate and Dopamine (NMDA/DA) interactions. The combined measures provide the opportunity to advance our understanding of specific aspects of brain function related to familial alcoholism vulnerability in an already well characterized population as some members evolve into alcohol abuse. In addition, as well as conventional within-task analyses, functional network connectivity and allied approaches will be used to examine brain networks across the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45 years
* Estimated full-scale IQ>70
* Individual can cooperate with all study procedures
* No history of neurological disorder (e.g., epilepsy)
* No major medical condition (e.g., cancer)
* No history of significant head trauma
* Stable medication treatment 6 weeks prior to study enrollment
* Negative urine drug and breathe alcohol test at time of MRI scan
* Negative urine pregnancy test at time of MRI scan
* No MR contra-indications (e.g., in-body metal implant, severe claustrophobia)
* No contra-indications to study drug

Exclusion Criteria:

* A diagnosis of any psychotic disorder, or current mood or anxiety disorders under DSM-V, using the SCID-V-RV psychiatric interview
* A current diagnosis of: a) Alcohol use disorder, if severe (AUD, mild or moderate OK if no craving, tolerance, and withdrawal 3 months prior to interview) b) Substance use disorder
* Report of psychotic disorder in a 1º relative
* Auditory or visual impairment that interferes with test-taking
* Prenatal exposure to alcohol plus currently meeting criteria for features of fetal alcohol syndrome
* Not speaking English fluently or being a non-native English speaker, or being educated in a primary language other than English > grade 1
* Intellectual Disability (Full Scale IQ<70)
* Traumatic brain injury with loss of consciousness > 30 minutes or concussion in last 30 days
* Presence or history of neurosurgery or any neurologic illness that may affect brain physiology (e.g., epilepsy, Multiple Sclerosis), including focal brain lesion seen on structural MRI (all structural scans are read by a board certified radiologist)
* A current major medical condition (e.g. cancer, heart failure)
* Current pregnancy (all females will be tested with urine screens on the day of MRI)
* Women not on an effective form of birth control/contraception or abstinent during time of study visits to prevent exposure of the investigational drug to suspected fetus
* Current substance use with the exception of marijuana (THC), provided last use of THC was 24+ hours before visit (All participants will receive a urine screen for the presence of marijuana, cocaine, opiates and a breath screen to detect the presence of alcohol)
* Inability to comprehend the consent form appropriately
* Inability to cooperate with study procedures
* Other specific fMRI exclusions include metal devices, clips or fragments in body (orbital xray performed if needed)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Nucleus accumbens (Nacc)/Ventral striatum (VS) BOLD activation during A1 phase in FHP on study medication vs. placebo | Mavoglurant and Placebo administration are 1 week apart
  Changes in NAcc/VS BOLD (Blood-oxygen-level-dependent) activation during the A1 loss anticipation prospect phase of the MRI Monetary Incentive Delay task in FHP while on mavoglurant compared to placebo
BOLD activation to alcohol vs. non-alcohol stimuli during ACR task alcohol versus non-alcohol stimuli | Mavoglurant and Placebo administration are 1 week apart
  Changes in BOLD response in FHP to alcohol versus non-alcohol stimuli in several brain clusters containing MFC, caudate, parahippocampal gyrus, temporal cortex and cerebellum, when administered mavoglurant compared to placebo

SECONDARY OUTCOMES:
Dynamic Causal Modeling (DCM)-determined relationships between nucleus accumbens (NAcc) and -medial PFC BOLD signal during MSDM task | Mavoglurant and Placebo administration are 1 week apart
  Dynamic Causal Modeling (DCM)-determined relationships between nucleus accumbens (NAcc) and -medial PFC BOLD signal during MSDM fMRI task in FHP while on mavoglurant compared to placebo
Regional differences in BOLD signal | Mavoglurant and Placebo administration are 1 week apart
  Impairment of top down inhibitory control and related cortical activation of the executive control network in FHP while on mavoglurant compared to placebo measured by regional differences in BOLD signaling

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey D Pearlson, MD, Principal Investigator — Yale University
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States